CLINICAL TRIAL: NCT02488213
Title: Effect of Nutritional Counseling Based on Diet Quality on Metabolic Control in Patients With Type 2 Diabetes Mellitus: Randomized Clinical Trial
Brief Title: Effect of Nutritional Counseling Based on Diet Quality on Metabolic Control in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-0585
Record Dates: First submitted 2015-03-09; First posted 2015-07-02 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Nutritional Counseling; Diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Diet Guidance (Active Comparator): The patients will receive usual diet guidance from the current nutritional recommendations for diabetes, according to the routine performed in outpatient patients treated in Endocrinology Division, Hospital de Clinicas de Porto Alegre.
  Interventions: Other: Usual Diet Guidance
- Nutritional Counseling (Experimental): The patients will receive nutritional counseling from the diet quality assessment with adopting some techniques of motivational interviewing, and delivery of educational support material.
  Interventions: Other: Nutritional Counseling

INTERVENTIONS:
Other: Nutritional Counseling — The patients with type 2 diabetes mellitus treated in Endocrinology Division, Hospital de Clinicas de Porto Alegre will receive nutritional counseling from the diet quality assessment with adopting some techniques of motivational interviewing, and delivery of educational support material. The patients will need to come to hospital for three more visits every two months throughout the study (2, 4, 6 months). They will also be contacted by telephone during the months when will not have query (1, 3 and 5 months). The study will total duration of six months.
  Arms: Nutritional Counseling
Other: Usual Diet Guidance — The patients with type 2 diabetes mellitus treated in Endocrinology Division, Hospital de Clinicas de Porto Alegre will receive usual diet guidance from the current nutritional recommendations for diabetes, according to the routine performed. The patients will need to come to hospital for three more visits every two months throughout the study (2, 4, 6 months). They will also be contacted by telephone during the months when will not have query (1, 3 and 5 months). The study will total duration of six months.
  Arms: Usual Diet Guidance

SUMMARY:
Randomized clinical trial with outpatient patients with type 2 diabetes mellitus treated in Endocrinology Division, Hospital de Clinicas de Porto Alegre. The study aims to carry out a nutritional counseling directed to offer benefits in metabolic control in diabetic patients.

DETAILED DESCRIPTION:
Randomized clinical trial with outpatient patients with type 2 diabetes mellitus treated in Endocrinology Division, Hospital de Clinicas de Porto Alegre. The study aims to carry out a nutritional counseling directed to offer benefits in metabolic control in diabetic patients. The initial step will be performed analysis of composition and diet quality, and anthropometric and laboratory evaluation. After initial assessment and meeting the criteria eligibility, patients will be randomized to receive nutritional counseling from diet quality (intervention group) or usual diet in according to current nutritional recommendations (control group). Both the groups will receive adjust caloric intake as the nutritional needs of each patient. Patients will be followed over six months, on a monthly basis from hospital visits or telephone monitoring. The outcomes evaluated will be: the achievement of therapeutic targets (fasting blood glucose levels between 70-130 mg / dL, HbA1c<7%, LDL cholesterol <100 mg/dL and triglycerides <150 mg/dL); use of antidiabetic drugs, lipid-lowering and antihypertensive drugs, and adherence to necessary dietary changes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients aged ≥ 30 years;
* Body mass index ≤ 40kg/m²;
* Serum creatinine <2 mg/dL;
* Serum triglycerides <400 mg/dL.

Exclusion Criteria:

* Cognitive impairment (clinical suspicion);
* Illiterate;
* Liver function tests and abnormal thyroid;
* Urinary tract infection carriers, kidney disease and heart failure uncompensated (grade III or IV);
* Active wasting disease diagnosis (Cancer, Acquired Immune Deficiency Syndrome);
* Metabolic control within the therapeutic target;
* Patients with dietary guidance by nutritionist in less than three months.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Glicemic control | six months
  Obtaining HbA1c <7% and/or reduction in HbA1c at least 1% of baseline

SECONDARY OUTCOMES:
Obtaining therapeutic target | six months
  Obtaining therapeutic target from laboratory evaluation: fasting blood glucose of 70 to 130mg/dL (serum measurement)
Obtaining therapeutic target | six months
  Obtaining therapeutic target from laboratory evaluation: LDL cholesterol <100mg/dL (serum measurement)
Obtaining therapeutic target | six months
  Obtaining therapeutic target from laboratory evaluation: triglycerides <150mg/dL (serum measurement)
Obtaining therapeutic target | six months
  Obtaining therapeutic target for average blood pressure <130/80 mmHg. There will be two measures separately, with one-minute interval, with the patient seated after five minutes of rest.
Adherence to nutritional counseling | six months
  Adherence to nutritional counseling will be measured from food surveys, telephone monitoring and implementation of a reliable scale to assess the degree of commitment to nutritional guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Jussara C de Almeida, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided